CLINICAL TRIAL: NCT05505578
Title: GamerFit: A Digital Intervention to Improve Physical Activity and Sleep Behaviors in Youth With Psychiatric Diagnoses
Brief Title: A Digital Intervention to Improve Physical Activity and Sleep Behaviors in Youth With Psychiatric Diagnoses
Acronym: GamerFit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Merrimack College (Other)
Responsible Party: Principal Investigator, Amanda Staiano, Associate Professor, Pennington Biomedical Research Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PBRC-2021-071
Record Dates: First submitted 2022-07-27; First posted 2022-08-17 (Actual); Results first posted 2025-05-01 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Psychiatric Diagnosis
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GamerFit Condition (Experimental): Includes use of a Fitbit and exergaming devices, the GamerFit app, and weekly telehealth coaching sessions.
  Interventions: Behavioral: GamerFit Condition
- Comparator Condition (Active Comparator): Youth assigned to the comparator condition (n=30-35) will receive a Fitbit device (same as the intervention condition) and the Fitbit account activated on their device (e.g. phone/tablet/computer). They will receive instructions on using the PA and sleep tracking features, as well as a booklet of healthy habit tips. They will receive reminders to charge, sync and review their Fitbit data for the duration of the intervention.
  Interventions: Behavioral: Comparator Condition

INTERVENTIONS:
Behavioral: GamerFit Condition — Participants receive a Fitbit device, the GamerFit app on their mobile device, exergaming console and games (Nintendo Switch) (where applicable), and follow a 12-week exergaming curriculum provided by the app. Physical activity (PA) increases during the intervention up to 60 minutes/session. Other interventional aspects include weekly reminders, exercise and health related video materials, and weekly telehealth sessions with an intervention coach.
  Arms: GamerFit Condition
Behavioral: Comparator Condition — Participants receive a Fitbit device, instructions on how to use it, and a booklet of healthy tips. They also get weekly reminders to charge, sync, and review their Fitbit data.
  Arms: Comparator Condition

SUMMARY:
The goal of "GamerFit" is to test the delivery of a theory-based mHealth app that utilizes social support, exergaming, and telehealth coaching to improve PA levels, sleep, and psychiatric symptoms among youth participants (ages 13-17 y) with PD. In order to aid future intervention optimization, up to 65 participants with at least one PD will be randomized, with 30-35 using the GamerFit app with weekly telehealth coaching sessions and 30-35 using a commercial healthy habits app as a comparator group

ELIGIBILITY:
Inclusion Criteria:

* 13-17 years of age (child/participant)
* At least one PD diagnosis (excluding eating disorders) confirmed by parent report of physician diagnosis (child/participant)
* IQ≥85/no intellectual disability that precludes participation confirmed by parent report (child/participant)
* Can understand verbal English-language exergaming instructions (child/participant)
* Physically capable of exercise confirmed by parent report (child/participant)
* Has access to a smart phone or compatible tablet (child/participant)
* Willing to download and use the app (child/participant)
* Willing and able to be present during telehealth coaching sessions (parent)
* Can have a competent translator present during coaching sessions if not fluent in English (parent)

Exclusion Criteria:

- Families for whom the mPIs think the study and/or intervention is clinically/medically inappropriate (e.g. developmental delay, or emotional or cognitive difficulties, if the PI believes these factors will interfere with study/intervention participation)

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 62 (Actual)
Dates: Start 2023-01-19 (Actual); Primary Completion 2024-03-12 (Actual); Study Completion 2024-03-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amanda E Staiano, PhD, MPP, Principal Investigator — Pennington Biomedical Research Center; April Bowling, MA, ScD, Principal Investigator — Merrimack College
Locations (2):
- United States (2):
  - Pennington Biomedical Research Center, Baton Rouge, Louisiana
  - Merrimack College, North Andover, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
Data will be made available to external investigators/public on a case-by-case basis, to be approved by the mPIs, in accordance with institutional, state, and federal regulations. All data that are shared will be de-identified to protect participant privacy and confidentiality. We will also make sure the data and relevant documents are available to users only under a data-sharing agreement that includes guarantees that: 1) data is used for research purposes only; 2) data will be secured on a password protected computer; and 3) data will be deleted after analyses are completed. Data and datasets will be kept and available to share for at least three years following completion of the project, in accordance with NIH regulations. Both institutions (Merrimack College and PBRC) have internal processes for data sharing and transfer lead by PBRC's Office of Legal and Regulatory Compliance and in accordance with the Office of Computing Services.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: December 2023 for 3 years

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | GamerFit Condition | Comparator Condition
Started | 31 | 31
Completed | 25 | 19
Not Completed | 6 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GamerFit Condition | Comparator Condition | Total
Number analyzed (Participants) | 31 | 31 | 62
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 31 | 31 | 62
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 7 | 15
  Male | 23 | 24 | 47
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 3 | 8
  Not Hispanic or Latino | 26 | 28 | 54
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 3 | 5
  White | 25 | 24 | 49
  More than one race | 3 | 3 | 6
  Unknown or Not Reported | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of the App
Description: Percentage of live coaching sessions attended (i.e. average of the number of coaching sessions attended divided by total number of coaching sessions expected). Because this is a percentage of visits, standard deviations/standard errors are not provided. This data are measured within the group as a whole and not by participants individually.
Time Frame: 12 weeks
Population: Participants randomized to the GamerFit group only received weekly telehealth sessions.
Measure: Number; unit: percentage of visits completed
Units Other Than Participants: Coaching Sessions
Arm/Group | GamerFit Condition
Number analyzed (Participants) | 31
Number analyzed (Coaching Sessions) | 12
percentage of visits completed | 88

2. Secondary Outcome: Physical Activity
Description: Change in average minutes of daily physical activity from baseline to 12 weeks (e.g. value at 12 weeks minus value at baseline).
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: minutes per day
Arm/Group | GamerFit Condition | Comparator Condition
Number analyzed (Participants) | 31 | 31
minutes per day | 20.12 (16.42) | 4.17 (18.63)

3. Secondary Outcome: Sleep
Description: Change in average minutes of daily sleep from baseline to 12 weeks (e.g. value at 12 weeks minus value at baseline).
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: minutes per day
Arm/Group | GamerFit Condition | Comparator Condition
Number analyzed (Participants) | 31 | 31
minutes per day | -6.5 (19.1) | 19.6 (21.4)

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | GamerFit Condition | Comparator Condition
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/31
Other Adverse Events (participants affected / at risk) | 0/31 | 0/31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-05-15): https://cdn.clinicaltrials.gov/large-docs/78/NCT05505578/Prot_SAP_000.pdf